CLINICAL TRIAL: NCT02351336
Title: Three - Dimensional Ultrasound Estimation of Fetal Adrenal Gland Enlargement Compared to Assessment of Cervical Changes Alone & Prediction of Impending Preterm Birth
Brief Title: Fetal Adrenal Gland Volume Estimation Compared to Cervical Length Assessment in Prediction of Preterm Birth
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wessam Magdy Abouelghar (Other)
Collaborators: Ain Shams Maternity Hospital (Other)
Responsible Party: Sponsor-Investigator, Wessam Magdy Abouelghar, Assisstant Professor of Obstetrics & Gynecology, Ain Shams Maternity Hospital
Organization: Ain Shams Maternity Hospital (Other)
Other Study IDs: PTB 012
Record Dates: First submitted 2015-01-22; First posted 2015-01-30 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Preterm Labour
Keywords: Threatened preterm birth; Fetal adrenal gland volume; Fetal zone enlargement; Prediction of preterm birth
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- threatened preterm labour: Women who are diagnosed as having threatened preterm labour based on the American college of obstetricians and gynaecologists guidelines (ACOG,2003) :
  * Presence of uterine contractions ( at least 4 in 20 minutes or 8 in 60 minutes )
  * Cervical dilataion >1cm, &/or
  * Cervical effacement ≥ 80%
  Interventions: Device: Ultrasound imaging

INTERVENTIONS:
Device: Ultrasound imaging — 1. - Fetal adrenal gland volume calculation using 3D ultrasound ( in mm3)
  2. - corrected adrenal gland volume calculation ( adrenal gland volume (mm3)/ estimated fetal weight (kg) )
  3. - CL measurement using 2D ultrasound ( in cm)

SUMMARY:
If the investigators could prove that three -dimensional ultrasound measurement of fetal adrenal gland volume can accurately predict the likelihood of preterm birth in patients having symptoms and signs of PTL , they would be able to use it as a valuable component for assessment and early management of high risk pregnant women for PTB which can be positively reflected on the risk of neonatal morbidity and mortality in those patients.

DETAILED DESCRIPTION:
Preterm birth ( PTB) is one of the leading causes of neonatal morbidity and mortality Early PTB (≤ 34 weeks' gestation) carries a 7-fold increased risk of Neonatal death . Following PTB, survivors can experience significant long term cognitive, behavioral, emotional, sensory, and motor deficits. Hence, there is growing interest in the identification of women who are at Risk for spontaneous PTB. Many biophysical and biochemical markers have been discovered to identify those women who are at risk for spontaneous PTB.

Unfortunately, none of the various maternal and fetal biomarkers such as:

cytokines, CRH, C-reactive protein, fetal fibronectin ,…. etc. are sufficiently sensitive or specific to be used alone or in combination to help decrease the rate of preterm births. Obviously, there's a need for an accurate method with high sensitivity and specificity for prediction of preterm labor. So that an appropriate management or referral to a higher center can be done to women likely to have PTB. Whereas unnecessary tocolytic therapy can be avoided in women who are unlikely to have PTB. Convincing data have shown that 2-dimensional (2D) ultrasound measurement of cervical length (CL) can identify women at risk for PTB.

Accordingly, CL is now widely used in clinical practice for risk estimation. However, as understanding of the mechanisms of preterm labor (PTL) have evolved, obstetricians have learned that, in some women, cervical shortening is a phenomenon that carries no increased risk for prematurity. Therefore, the search for early and accurate markers that distinguish between physiologic processes and abnormal activation of the labor cascade has been ongoing.

Literature has suggested that activation of the fetal hypothalamic-pituitary-adrenal axis play a crucial rule in commencement of labor. A previous study demonstrated that three -dimensional ultrasound measurement of fetal adrenal gland volume (AGV) may identify women at risk for impending PTB. In a more recent study receiver operator characteristics (ROC) curve analysis revealed that three -dimensional ultrasound measurement of (AGV) was superior to two-dimensional ultrasound measurement of (AGV) for anticipation of PTB within 7 days of the scan. The aim of this study is to investigate the utility of 3D fetal adrenal gland volume measurement in the early prediction of PTB and to determine whether these measurements could be combined with 2D ultrasound cervical assessment to improve the early prediction of PTB.

ELIGIBILITY:
Inclusion Criteria:

1. Age : 18 - 40 years
2. Gestational age: 26 - 35 weeks , which is going to be calculated according to the date of last menstrual period & confirmed by first trimester ultrasonography .
3. Women who are diagnosed as having threatened preterm labour based on the American college of obstetricians and gynaecologists guidelines (ACOG,2003) :

   * Presence of uterine contractions ( at least 4 in 20 minutes or 8 in 60 minutes )
   * Cervical dilataion >1cm, &/or
   * Cervical effacement ≥ 80% 4. Women having one or more of the following:

     * Multifetal pregnancy .
     * Previous preterm labor or premature birth, particularly in the most recent pregnancy or in more than one previous pregnancy

Exclusion Criteria:

1. Suspected fetal growth restriction .
2. Preterm premature rupture of the membranes : confirmed by visualization of amniotic fluid vaginal pooling at the time of sterile speculum examination .
3. Patients with antepartum haemorrhage ( due to placental abruption &/or placenta previa )
4. Presence of fetal anomalies incompatible with life. 5 - Patients who are not sure of dates

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who are diagnosed as having threatened preterm labour based on the American college of obstetricians and gynaecologists guidelines (ACOG,2003) :
  * Presence of uterine contractions ( at least 4 in 20 minutes or 8 in 60 minutes )
  * Cervical dilataion >1cm, &/or
  * Cervical effacement ≥ 80%
Sampling Method: Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
1. Accurate prediction of impending preterm birth using 3D ultrasound estimation of fetal adrenal gland volume | within 7 days of ultrasound scan

SECONDARY OUTCOMES:
Superiority of Adrenal gland volme estimation in prediction of preterm birth compared to cervical length measurement alone | 7 days of ultrasound scan

CONTACTS AND LOCATIONS:
Overall Officials: Wessam M Abouelghar, MD, Study Director — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

REFERENCES:
- [Background] Turan OM, Turan S, Funai EF, Buhimschi IA, Campbell CH, Bahtiyar OM, Harman CR, Copel JA, Buhimschi CS, Baschat AA. Ultrasound measurement of fetal adrenal gland enlargement: an accurate predictor of preterm birth. Am J Obstet Gynecol. 2011 Apr;204(4):311.e1-10. doi: 10.1016/j.ajog.2010.11.034. Epub 2011 Feb 3. PMID 21292230
- See also: Ultrasound measurement of fetal adrenal gland enlargement: an accurate predictor of preterm birth. — http://www.ncbi.nlm.nih.gov/pubmed/21292230